CLINICAL TRIAL: NCT05858203
Title: Inhibition of Che-1/AATF as a New Tool in Multiple Myeloma Treatment
Acronym: AATF/Che-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS1442/20
Record Dates: First submitted 2023-03-24; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Chromatin Immunoprecipitation Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ATAC-seq and ChIP-seq — CD138+ cells will be isolated from the bone marrow of MM patients and will be subjected to ATAC-seq and ChIP-seq analyses, by useing specific antibodies, to better understand the involvment of Che-1 in MM tumorogenesis.

SUMMARY:
Multiple myeloma (MM) is a haematological malignancy characterized by the accumulation of proliferating antibody producing plasma cells in the bone marrow. In the last few years many studies have emphasized the biological complexity and heterogeneity of MM as a result of both genetic and epigenetic aberrations. Che-1/AATF (Che-1) is a transcriptional cofactor involved in cell cycle regulation, apoptosis, DNA damage and stress response. it can be hypothesized that Che-1 might contribute to the establishment of the MM malignant phenotype by sustaining global transcription through its ability to modulate chromatin accessibility.

The prospective study on MM human samples aims to understand the involvement of Che-1 in the transcriptional regulation and chromatin remodeling during the pathology. To this goal the main objectives are:

* Characterization of Che-1's role in chromatin remodeling and global gene expression
* Study in vivo and in vitro of Che-1 involvement in MM tumorigenesis
* Evaluation of Che-1 as a possible therapeutic target

ELIGIBILITY:
Inclusion Criteria:

* MM Patients

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MM Patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Che-1 involvement in MM tumorigenesis | About 2 years
  Characterization of Che-1's role in chromatin remodeling and global gene expression

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Regina elena Cancer Institute, Roma
  - "Regina Elena" National Cancer Institute, Rome